CLINICAL TRIAL: NCT04590118
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of a Multicenter, Blind, Randomized, Placebo Controlled Single Injection of It-hMSC in Patients With Ischemic Stroke
Brief Title: Allogeneic Mesenchymal Stem Cells for the Survivors of Ischemic Stroke Trial (ASSIST)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiuzhitang Maker (Beijing) Cell Technology Co.,Ltd. (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STCMSC-CT-001
Record Dates: First submitted 2020-09-07; First posted 2020-10-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: In phase I, the masking method is open-label, whereas in phase II, the masking method is double blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: it-hMSC (Experimental): Single intravenous infusion of 0.5×10^6, 1×10^6, 2×10^6 it-hMSC/kg
  Interventions: Drug: it-hMSC
- Placebo-controlled: Placebo (Placebo Comparator): Single intravenous infusion of 1 ml/kg placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: it-hMSC — Single intravenous infusion of it-hMSC for ischemic stroke patients
  Arms: Experimental: it-hMSC
Drug: Placebo — Single intravenous infusion of 1 ml/kg placebo
  Arms: Placebo-controlled: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary efficacy of single injection of it-hMSC in patients with ischemic stroke in a multicenter, blind, randomized, placebo controlled trial

DETAILED DESCRIPTION:
Stroke is a leading cause of disability. According to the comprehensive standardized prevalence estimation in 2016, 12.42 million people older than 40 years in China are currently suffering from stroke or have ever suffered from stroke. The overall prevalence rate of stroke in China was 1,596 per 100,000 people in 2016, 4.6 times higher than the rate of 345.1 per 100,000 people in 2013 and 70% of the survivors have disabilities in varying degrees. In addition to rehabilitation therapy, there is no therapeutic drugs of remarkable curative effect for the treatment of ischemic stroke patients. The latest data show that the annual recurrence rate of ischemic stroke in China is as high as 17.7%.

Allogeneic mesenchymal stem cells have been used in many clinical studies for different diseases. In addition to differentiating into multiple cell types and promoting the recovery and repair of the brain by replacing damaged cells, mesenchymal stem cells also secrete cytokines and neurotrophic factors to support and stimulate the growth of other endogenous cells. Meanwhile, mesenchymal stem cells also have anti-inflammatory and immunomodulatory functions. These characteristics of mesenchymal stem cells provide a new therapy for the treatment of stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Clinical diagnosis of ischemic stroke for more than 6 months.
* Imaging findings suggestive of ischemic stroke with functional deficits at initial diagnosis and enrollment.
* Severe neurological impairment associated with the diagnosis of ischemic stroke that resulted in the subject needing assistance to walk or not being able to perform general daily activities independently.
* No substantial improvement in neurologic or functional deficits for the 2 months prior to enrollment.
* NIHSS score between 6-20.
* Life expectancy longer than 12 months.
* Prior to treatment, the patient received standard medical care for secondary prevention of ischemic stroke, including but not limited to appropriate blood pressure and cholesterol control measures, use of antiplatelet agents or anticoagulants (except when prohibited).
* Understand and provide signed informed consent, or have a designated legal guardian or spouse make such decision voluntarily on behalf of the subject.
* Expected that the patient will receive standard medical care for secondary prevention of ischemic stroke and participate in all planned safe follow-up visits reasonably.
* Organ function as defined by the following criteria:

AST ≤ 2.5×ULN ALT ≤ 2.5×ULN TSB ≤1.5×ULN PT ≤1.25×ULN and PTT ≤1.25×ULN in subjects who did not receive antithrombotic therapy Serum albumin ≥ 3.0g/dL ANC ≥ 1,500/μL Platelets ≥ 150,000/μL Hemoglobin ≥ 9.0g/dL Serum creatinine ≤ 1.5×ULN Serum amylase or lipase ≤ 1.0×ULN

Exclusion Criteria:

* History of epilepsy.
* History of cancer.
* History of brain trauma and brain tumor.
* Positive for hepatitis B surface antigen, E antigen, E antibody, core antibody, hepatitis C, HIV or RPR.
* Myocardial infarction occurred within six months of study entry.
* Any other medical problems of clinical significance, abnormal mental or test results that the investigator or sponsor determined participating in the study pose a safety risk to the subject.
* Imaging findings suggestive of subarachnoid hemorrhage or intracerebral hemorrhage in the past 12 months.
* Participation in any study of experimental drug or device within 3 months.
* Participation in other study related to stem cell-therapy.
* History of drug or alcohol abuse within 1 year.
* Pregnant, lactating or planning to become pregnant during the trial.
* Allergic to cattle or pork products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events assessed by CTCAE V5.0 during the twelve-month study period after it-hMSC infusion. | 12 months

SECONDARY OUTCOMES:
Modified Rankin Scale | month 1, month 3, month 6, month 9, month 12
  The change from the baseline in Modified Rankin Scale will be calculated at month 1, month 3, month 6, month 9, month 12 post-treatment, as available.
  The scale is divided into 7 degrees, from 0 (no deficit) to 6 (dead).
National Institute of Health stroke scale | month 1, month 3, month 6, month 9, month 12
  The change from the baseline in National Institute of Health stroke scale will be calculated at month 1, month 3, month 6, month 9, month 12 post-treatment, as available.
  The range of scores is from 0 (normal) to 42.
Mini-mental State Examination | month 1, month 3, month 6, month 9, month 12
  The change from the baseline in Mini-mental State Examination will be calculated at month 1, month 3, month 6, month 9, month 12 post-treatment, as available.
  The range of scores is from 0 to 30 (normal).
Barthel Index | month 1, month 3, month 6, month 9, month 12
  The change from the baseline in Barthel Index will be calculated at month 1, month 3, month 6, month 9, month 12 post-treatment, as available.
  The range of scores is from 0 to 100 (normal).
Geriatric Depression Scale | month 1, month 3, month 6, month 9, month 12
  The change from the baseline in Geriatric Depression Scale will be calculated at month 1, month 3, month 6, month 9, month 12 post-treatment, as available.
  The range of scores is from 0 (normal) to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China